CLINICAL TRIAL: NCT01848314
Title: The Effect of Renal Denervation on Renal Flow in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, W.I. Verloop, MD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NL42766.041.12
Record Dates: First submitted 2013-04-26; First posted 2013-05-07 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing renal denervation (Experimental): patients diagnosed with resistant hypertension, eligible to undergo renal denervation
  Interventions: Procedure: Renal Denervation

INTERVENTIONS:
Procedure: Renal Denervation — Flowmeasurements will be performed before and after renal denervation
  Other Names: flowmeasurements

SUMMARY:
Many studies have studied the effect and safety of renal denervation. However, it remains unknown what the exact mechanism behind renal denervation is. It can be hypothesized that a difference in renal blood flow occurs after treatment. In the light of this ignorance, current study will investigate whether renal denervation leads to a difference in renal blood flow after treatment with renal denervation.

ELIGIBILITY:
Inclusion Criteria:

* Individual is scheduled to undergo renal denervation as standard patient care for resistant hypertension.
* Individual is diagnosed with resistant hypertension. Secondary causes and a white coat hypertension are actively excluded.
* Individual is ≥18 years of age.
* Individual agrees to have all study procedures performed, and is competent and willing to provide written informed consent to participate in this clinical study.

Exclusion Criteria:

* Individual is excluded from treatment with pRDN .
* Individual has an estimated glomerular filtration rate (eGFR) of <30mL/min/1.73m2, using the MDRD calculation.
* Individual has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months of the screening visit, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
* Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, haemophilia or significant anaemia).
* Individual is pregnant, nursing or planning to be pregnant.
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in microvascular resistance | Within 30 minutes after renal denervation

SECONDARY OUTCOMES:
change in average flow velocity | within 30 minutes after renal denervation

OTHER OUTCOMES:
safety of measurement | within 24 hour after renal denervation

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Voskuil, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands